CLINICAL TRIAL: NCT05752162
Title: Perioperative Complications Linked to COVID-19 History in Elective Cardiac Surgery Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Cornelia Elena Predoi, phD student, Carol Davila University of Medicine and Pharmacy
Other Study IDs: 20083/11.07.2022
Record Dates: First submitted 2023-02-28; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Complications; COVID-19
MeSH Terms: conditions — Postoperative Complications; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A. Primary objective

Identifying risk factors for peri-operative complications in patients who have had COVID-19.

B. Secondary objectives

Identifying peri-operative complications in patients who have had COVID-19. Follow-up of peri-operative complications during hospitalization. Identifying the safe distance at which a patient can be operated after a Sars CoV2 infection without having an increased risk of peri-operative complications.

C. Study inclusion and exclusion criteria

1. Inclusion criteria

   Patients should be included if:
   * are scheduled for elective cardiac surgery with extracorporeal circulation (bypass);
   * they give their consent for their data to be included in studies;
2. Exclusion criteria

Patients should be excluded if:

* they have emergency surgery;
* have had Sars Cov 2 infection more recently than 3 months;

D. Data Collection

It is done in an excel table. Data collection is done anonymously. No patient-identifying data will be collected. The collected data will be about comorbidities, COVID-19 status - disease and vaccination, postoperative complications.

DETAILED DESCRIPTION:
Types of data collection from the patients:

The type of surgery Age Sex Smoking Diabetes History of renal disease Preoperative anemia Preoperative creatinine Preoperative urea BMI NYHA class ASA score EuroScore I Preoperative LVEF Disease COVID -19 Date of illness Hospitalization for COVID-19 COVID 19 vaccination status Necessary vasopressor peri-operative duration and Maximum dose Perioperative positive inotrope required Bypass duration Duration of Aortic clamping Intraoperative transfusions Post operative creatinine - peak level Post-operative urea peak level Duration of post-operative oro-tracheal intubation NIV required Duration of hospitalization in Cardiac Intensive Care Unit Duration of postoperative hospitalization

ELIGIBILITY:
Inclusion Criteria:

* are scheduled for elective cardiac surgery with extracorporeal circulation (bypass);
* they give their consent for their data to be included in studies;

Exclusion Criteria:

* they have emergency surgery;
* have had Sars Cov 2 infection more recently than 3 months;

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in the Cardiac Intensive Care Unit 2 IUBCV CC Iliescu for postoperative management.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Identifying risk factors for peri-operative complications in patients who have had COVID-19 | 3 years

SECONDARY OUTCOMES:
Identifying peri-operative complications in patients who have had COVID-19 | 3 years
  Follow-up of peri-operative complications during hospitalization.
Identifying the safe distance at which a patient can be operated after a Sars CoV2 infection without having an increased risk of peri-operative complications. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- IUBCV Prof. Dr. CC Iliescu, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] COVIDSurg Collaborative. Outcomes and Their State-level Variation in Patients Undergoing Surgery With Perioperative SARS-CoV-2 Infection in the USA: A Prospective Multicenter Study. Ann Surg. 2022 Feb 1;275(2):247-251. doi: 10.1097/SLA.0000000000005310. PMID 34793350
- [Result] Wajekar AS, Solanki SL, Divatia JV. Pre-Anesthesia Re-Evaluation in Post COVID-19 Patients Posted for Elective Surgeries: an Online, Cross-Sectional Survey. Indian J Surg Oncol. 2021 Dec;12(Suppl 2):234-239. doi: 10.1007/s13193-021-01347-z. Epub 2021 May 17. PMID 34025062